CLINICAL TRIAL: NCT03755830
Title: Study of the Cutaneous Expression of Prostaglandin F2-alpha (PGF2α) in Vitiligo Patients: a Case-control Study.
Brief Title: Prostaglandin F2-alpha (PGF2α) in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dermatology 10
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitiligo patients (Active Comparator): Two skin biopsies (lesional and non-lesional) will be taken from every patient.
  Interventions: Other: Skin biopsy
- healthy controls (Experimental): A skin biopsy will be taken from each control subject.
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — Two skin biopsies (lesional and non-lesional) will be taken from every patient. Also a skin biopsy will be taken from each control subject.

SUMMARY:
study the cutaneous expression of PGF2α in vitiligo patients and compare it with normal control subjects.

DETAILED DESCRIPTION:
Measurement of tissue levels of PGF2α in vitiligo patients and compare them with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo.
* Both sexes.
* Age < 18 years old.
* New cases or cases not receiving any medications for at least 3 months ago.

Exclusion Criteria:

* Age: Patients < 18 years.
* Segmental or universal vitiligo.
* Pregnant and lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of tissue levels of PGF2α in vitiligo patients and compare them with healthy controls. | 6 months
  Measurement of tissue levels of PGF2α in vitiligo patients and compare them with healthy controls to study and verify the hypothesis of involvement of PGF2α in the pathogenesis of vitiligo.• Skin biopsy for assessment of tissue levels of the PGF2α will be taken from both lesional and non lesional skin of patients of vitiligo and from normal skin of healthy controls. All skin biopsies are from non-sun exposed sites.